CLINICAL TRIAL: NCT02383979
Title: Perioperative Visual Therapy May Help Prevent Phantom Limb Pain
Brief Title: Perioperative Mirror Therapy and Phantom Limb Pain
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NMCSD.2010.0007
Record Dates: First submitted 2015-03-04; First posted 2015-03-10 (Estimated); Last update posted 2019-08-28 (Actual); Status verified 2019-08

CONDITIONS: Phantom Limb Pain; Phantom Pain; Phantom Sensation; Pseudomelia
Keywords: Phantom limb pain; Mirror therapy; Elective amputation; Residual limb pain; Functional MRI
MeSH Terms: conditions — Phantom Limb | interventions — Mirror Movement Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Plasma Ball (Control) (Sham Comparator): Subjects randomized to standard therapy will participate 14 days of daily mirror therapy sessions preoperatively which will consist of undergoing a sham therapy with a 22" plasma globe involving contralateral limb interaction with the sphere.
  Interventions: Device: Sham (Comparator) Plasma Ball
- Experimental (Experimental): Subjects randomized to the mirror therapy limb will undergo 14 days of daily mirror therapy sessions preoperatively which will consist of observing the unaffected limb reflected for 30 minutes in a mirror positioned in the midline to block the view of the affected limb.
  Interventions: Device: Mirror
- Non-Surgical (No Intervention): Subjects will undergo 3 questionnaires and one functional fMRI exam. Imaging protocol will be identical to preoperative imaging protocol for amputation subjects. This data will aid in establishing baseline fMR activation values for all fMR paradigms tested. The control group will not be randomized to receive either perioperative plasma ball (sham) or mirror therapy.

INTERVENTIONS:
Device: Sham (Comparator) Plasma Ball — will consist of undergoing a sham therapy with a 22" plasma globe involving contralateral limb interaction with the sphere.
  Arms: Plasma Ball (Control)
Device: Mirror — will undergo 14 days of daily mirror therapy sessions preoperatively which will consist of observing the unaffected limb reflected for 30 minutes in a mirror positioned in the midline to block the view of the affected limb
  Arms: Experimental

SUMMARY:
Mirror therapy will consist of observing the unaffected limb reflected in a mirror positioned in the midline to block the view of the affected limb. All therapy sessions will be supervised by a physical therapist with the exception of weekends when the patients will continue therapy on an independent basis. In an effort to objectively demonstrate cortical reorganization associated with mirror therapy, patients can elect to participate in a functional MRI (fMRI) portion of the study. The fMRI would be evaluated prior to initiating the experimental or control therapy (Due to the sensitive timeline in this population and its effect on recruitment, we have amended the protocol to allow recruitment and enrollment to take place even if the timeline does not allow for the fMRI to be executed 2 weeks prior to amputation. Though this would be ideal, we will accept subjects that are only available for day before amputation scans), just before the operative procedure, at four weeks post-operation and then again at one year. All subjects will be evaluated at 4 weeks, 8 weeks (functional physical therapy (PT) tests only) 12 weeks, and 12 months postoperatively to determine 1) the incidence, severity and functional impact of phantom limb pain 2)the ability to meet various specialists' endpoints, to include participation in physical therapy, and 3) overall quality of life which the patients can describe subjectively. This therapy could have a dramatic impact on the long term prognosis of amputees whether due to trauma, metabolic conditions, tumor, or peripheral vascular disease.

This protocol will include performing fMRIs on a cohort of healthy, active duty, age matched, male personnel to create reference data to compare the fMRI data of study participants.

DETAILED DESCRIPTION:
Subjects scheduled for amputation will be randomized to either receive perioperative plasma ball (sham) or mirror therapy, which involves a daily session of 30 minutes of performing physical therapy exercises using either a mirror or plasma ball under the supervision of a certified physical therapist. Subjects scheduled to undergo limb amputation who opt in for the fMRI portion of the study will undergo a pre-treatment baseline fMRI (2 weeks prior to scheduled amputation, if possible, but as late as 1 day pre-operative), a post-mirror or sham therapy (preoperative-day before) fMRI, post-operative fMRI at 4 weeks and one year. Performing a baseline fMRI prior to any treatment, will provide objective data regarding the location and extent of cortical involvement prior to initiating mirror therapy. Those subjects randomized to the mirror therapy limb will undergo 14 days of daily mirror therapy sessions preoperatively which will consist of observing the unaffected limb reflected for 30 minutes in a mirror positioned in the midline to block the view of the affected limb. Those randomized to standard therapy will participate in an equivalent period of time undergoing a sham therapy with a 22" plasma globe involving contralateral limb interaction with the sphere. All therapy sessions will be supervised by a physical therapist with the exception of weekends when the patients will continue therapy on an independent basis. The subjects will then undergo a repeat fMRI (or first baseline, depending if pre-operative fMRI was possible) after completion of preoperative mirror or sham therapies and prior to surgical amputation to evaluate for changes suggestive of mirror therapy induced normalization in cortical patterns.

Control subject group will undergo 3 questionnaires and one functional fMRI exam. Imaging protocol will be identical to preoperative imaging protocol for amputation subjects. This data will aid in establishing baseline fMR activation values for all fMR paradigms tested. The control group will not be randomized to receive either perioperative plasma ball (sham) or mirror therapy.

All Subjects scheduled for surgery will then undergo amputation under the anesthetic technique of provider choice. If regional/neuraxial anesthetic techniques are used they will be standardized up to 1 day preoperative and 3 days postoperative. If using dexmedetomidine and/or ketamine infusions, their use will be limit to intraoperative periods at doses of 0.2 mcg/kg/hr and 0.15mg/kg/hr limit respectively. Anesthesiologist/Anesthetist choice will be permitted for all other intraoperative and postoperative meds. Within 1 week of amputation subjects will again repeat 14 days of their respectively assigned therapy limbs as described above in addition to routine post amputation care. All subjects will then be evaluated at four weeks postoperatively with measures delineated in section 5.(Statistics) to determine 1) incidence and severity of phantom limb pain 2) participation in therapy and ability to meet functional endpoints 3) quality of life. These same measures will be assessed at 12 weeks (3 months) and again at one year post procedure. A repeat fMRI will be obtained in those Subjects participating in the fMRI limb in order to evaluate how the postoperative cortical mapping compares to prior preoperative and postoperative studies.

ELIGIBILITY:
Inclusion Criteria:

Treatment (Surgical) Group:

1. Subjects age 18 years or older scheduled for elective amputation;
2. Cooperative, patient scheduled for amputation, with time and availability to do fMRI prior to their operative date;
3. Willing to perform mirror therapy for 14 days prior and post-operative procedure;
4. Subjects who opt for fMRI portion of the study are willing and/or able to tolerate fMRI.

Control (Non-Surgical) Group:

1. Subjects age 18 years to 30;
2. who are non amputated and healthy;
3. Cooperative, with time and availability to do an fMRI;
4. Willing and able to tolerate fMRI.

Exclusion Criteria:

1. inability to cooperate with physical therapy; and
2. possessing a contraindication to mirror therapy for example blindness or inability to position properly for the therapy
3. primary central nervous disease such as status post cerebral vascular accident with persistent deficit, Alzheimer's disease or Multiple Sclerosis. In addition, patients with claustrophobia will be excluded from participating in the fMRI portion of this study.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 115 (Estimated)
Dates: Start 2010-08; Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Comparing fMRI scans to see if mirror therapy helps prevent or alleviate phantom limb pain in service members undergoing amputation(s) | 4 weeks prior to surgery through 1 year post operation
  For patients participating in the fMRI procedures, the scans will be compared among the four time-points (pre-initiation of mirror therapy (if possible), post-mirror therapy but pre-amputation, post-amputation at 4 weeks and at one year post-amputation). Primary analysis will compare the two treatment groups from baseline to 4 weeks following the initial catheter placement; but additional comparisons will be completed to help plan future investigations.

CONTACTS AND LOCATIONS:
Overall Officials: Steven R Hanling, MD, Principal Investigator — United States Naval Medical Center, San Diego
Locations (1):
- Pain Medicine Center, Department of Anesthesiology, Naval Medical Center San Diego, San Diego, California, United States

REFERENCES:
- [Background] Mishra S, Bhatnagar S, Gupta D, Diwedi A. Incidence and management of phantom limb pain according to World Health Organization analgesic ladder in amputees of malignant origin. Am J Hosp Palliat Care. 2007 Dec-2008 Jan;24(6):455-62. doi: 10.1177/1049909107304558. Epub 2007 Sep 21. PMID 17890346
- [Background] Ramachandran VS, Hirstein W. The perception of phantom limbs. The D. O. Hebb lecture. Brain. 1998 Sep;121 ( Pt 9):1603-30. doi: 10.1093/brain/121.9.1603. PMID 9762952
- [Background] Flor H, Birbaumer N. Phantom limb pain: cortical plasticity and novel therapeutic approaches. Curr Opin Anaesthesiol. 2000 Oct;13(5):561-4. doi: 10.1097/00001503-200010000-00013. PMID 17016358
- [Background] Arnstein PM. The neuroplastic phenomenon: a physiologic link between chronic pain and learning. J Neurosci Nurs. 1997 Jun;29(3):179-86. doi: 10.1097/01376517-199706000-00005. PMID 9220365
- [Background] Ramachandran VS, Rogers-Ramachandran D. Synaesthesia in phantom limbs induced with mirrors. Proc Biol Sci. 1996 Apr 22;263(1369):377-86. doi: 10.1098/rspb.1996.0058. PMID 8637922
- [Background] Mercier C, Reilly KT, Vargas CD, Aballea A, Sirigu A. Mapping phantom movement representations in the motor cortex of amputees. Brain. 2006 Aug;129(Pt 8):2202-10. doi: 10.1093/brain/awl180. Epub 2006 Jul 14. PMID 16844715
- [Background] MacIver K, Lloyd DM, Kelly S, Roberts N, Nurmikko T. Phantom limb pain, cortical reorganization and the therapeutic effect of mental imagery. Brain. 2008 Aug;131(Pt 8):2181-91. doi: 10.1093/brain/awn124. Epub 2008 Jun 20. PMID 18567624
- [Background] Birbaumer N, Lutzenberger W, Montoya P, Larbig W, Unertl K, Topfner S, Grodd W, Taub E, Flor H. Effects of regional anesthesia on phantom limb pain are mirrored in changes in cortical reorganization. J Neurosci. 1997 Jul 15;17(14):5503-8. doi: 10.1523/JNEUROSCI.17-14-05503.1997. PMID 9204932
- [Background] Liepert J, Bauder H, Wolfgang HR, Miltner WH, Taub E, Weiller C. Treatment-induced cortical reorganization after stroke in humans. Stroke. 2000 Jun;31(6):1210-6. doi: 10.1161/01.str.31.6.1210. PMID 10835434
- [Background] Sterr A, Elbert, T, Rostroh B. Functional reorganization of human cerebral cortex and its perceptual concomitants. In: Fahle M, Poggio T. Terceptual Learning. MIT Press, 2002: 138.
- [Background] Jensen TS, Krebs B, Nielsen J, Rasmussen P. Phantom limb, phantom pain and stump pain in amputees during the first 6 months following limb amputation. Pain. 1983 Nov;17(3):243-256. doi: 10.1016/0304-3959(83)90097-0. PMID 6657285
- [Background] Dworkin RH, Turk DC, Farrar JT, Haythornthwaite JA, Jensen MP, Katz NP, Kerns RD, Stucki G, Allen RR, Bellamy N, Carr DB, Chandler J, Cowan P, Dionne R, Galer BS, Hertz S, Jadad AR, Kramer LD, Manning DC, Martin S, McCormick CG, McDermott MP, McGrath P, Quessy S, Rappaport BA, Robbins W, Robinson JP, Rothman M, Royal MA, Simon L, Stauffer JW, Stein W, Tollett J, Wernicke J, Witter J; IMMPACT. Core outcome measures for chronic pain clinical trials: IMMPACT recommendations. Pain. 2005 Jan;113(1-2):9-19. doi: 10.1016/j.pain.2004.09.012. No abstract available. PMID 15621359
- [Background] Farrar JT, Young JP Jr, LaMoreaux L, Werth JL, Poole MR. Clinical importance of changes in chronic pain intensity measured on an 11-point numerical pain rating scale. Pain. 2001 Nov;94(2):149-158. doi: 10.1016/S0304-3959(01)00349-9. PMID 11690728
- [Background] Cleeland CS, Ryan KM. Pain assessment: global use of the Brief Pain Inventory. Ann Acad Med Singap. 1994 Mar;23(2):129-38. PMID 8080219
- [Background] Cleeland CS, Nakamura Y, Mendoza TR, Edwards KR, Douglas J, Serlin RC. Dimensions of the impact of cancer pain in a four country sample: new information from multidimensional scaling. Pain. 1996 Oct;67(2-3):267-73. doi: 10.1016/0304-3959(96)03131-4. PMID 8951920
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Fischer, J: United States Military Casualty Statistics: Operation Iraqi Freedom and Operation Enduring Freedom. Congressional Research Service. March 25, 2009
- [Background] Chan BL, Witt R, Charrow AP, Magee A, Howard R, Pasquina PF, Heilman KM, Tsao JW. Mirror therapy for phantom limb pain. N Engl J Med. 2007 Nov 22;357(21):2206-7. doi: 10.1056/NEJMc071927. No abstract available. PMID 18032777